CLINICAL TRIAL: NCT03502915
Title: Randomized Controlled Trial of Nitrous Oxide Analgesia in External Cephalic Version (ECV)
Brief Title: Nitrous Oxide for External Cephalic Version
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-1569
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-03

CONDITIONS: External Cephalic Version
Keywords: breech presentation; nitrous oxide; analgesia; pregnancy
MeSH Terms: conditions — Breech Presentation; Agnosia | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Nitronox device will be covered. The person setting up the device with either 100% oxygen or 50% nitrous/50% oxygen, will not be participating in the study. The patient, investigator and labor and delivery personnel (obstetrician and nursing staff) will be blinded as to the medication being administered during the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nitrous Oxide (Experimental): Patients will receive nitrous oxide during the version procedure.
  Interventions: Drug: Nitrous Oxide
- Oxygen (Placebo Comparator): Patients will receive placebo (100% oxygen) during the version procedure.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nitrous Oxide — 50% nitrous oxide/50% oxygen via Nitronox delivery device
  Other Names: Laughing gas
  Arms: Nitrous Oxide
Other: Placebo — 100% oxygen via Nitronox delivery device
  Arms: Oxygen

SUMMARY:
This study seeks to determine the effectiveness of nitrous oxide in reducing the anxiety and pain associated with external cephalic version (ECV); a maneuver to turn the fetus from breech to cephalic position.

DETAILED DESCRIPTION:
Study Procedures:

Potential subjects will be identified as they are scheduled to undergo ECV at the UNC Department of Obstetrics and Gynecology. Subjects will be enrolled in the study by one of the study investigators. Details of the study will be reviewed with potential subjects and those wishing to enroll in the study will be consented for the study by one of the study investigators. Once enrolled participants will be randomized to receive either a mixture of 50% nitrous oxide in 50% oxygen or 100% oxygen, both of which will be delivered via the Nitronox apparatus. Demographic variables will be recorded for each participant at the time they are enrolled in the study

The Nitronox apparatus will be set up to deliver either 50% nitrous oxide in 50% oxygen or 100% oxygen by an anesthesia provider covering labor and delivery who is not involved in the study. The Nitronox device will be covered to prevent participants, study investigators and obstetricians performing the procedure from knowing whether nitrous oxide is being delivered. Nitrous oxide is odorless and colorless, so in that way is indistinguishable from oxygen.

Participants will be prepared for ECV according to current protocols for ECV at UNC. IV access will be obtained and tocolytic agents will be given according to current practice and protocols. Monitoring of maternal and fetal vital signs will be done according to current protocols.

Immediately before an ECV attempt participants will breathe through the facemask of the Nitronox device for 30 seconds and will then be free to use the device ad lib during the ECV attempt. Immediately following each attempt, while fetal monitoring is occurring, the participants will be asked to rate their maximum pain score during the previous attempt. They will also be asked to rate their current level of anxiety. This process will be repeated for any further ECV attempts.

At conclusion of all ECV attempts, while fetal monitoring is occurring, the participants will be asked to rate their current level of pain, their satisfaction with the procedure and about any side effects they experienced (nausea, vomiting, dizziness, headache, other). Participants will continue to be monitored on labor and delivery as current protocol dictates, typically 30 minutes of maternal and fetal monitoring if there are no complications and fetal status is reassuring.

Following the procedure, the obstetrician who performed the procedure will be asked to rate how difficult they felt it was to perform the procedure and to rate how much they felt the analgesic provided assisted in performing the procedure. They will also be asked to indicate whether they thought the patient was in the treatment or placebo arm of the study. This will be recorded to address the adequacy of blinding.

All study variables will be assessed and recorded by one of the study investigators to ensure consistency in data collection.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years or greater
* Scheduled to undergo external cephalic version due to singleton breech presentation
* Not scheduled to have spinal or epidural anesthesia during the version procedure
* American Society of Anesthesiology (ASA) Physical Status 1, 2 or 3.
* Able to provide informed consent and adhere to study protocol

Exclusion Criteria:

* Current or historical evidence of any clinically significant disease or condition, especially cardiovascular or neurological conditions that, in the opinion of the Investigator, may increase the risk of exposure to nitrous oxide or complicate the subject's post-procedural course.
* Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females will participate because only females can be pregnant.
Enrollment: 48 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A. Smith, MD, FASA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 9-36 months after publication
Access Criteria: Approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Hannah ME, Hannah WJ, Hewson SA, Hodnett ED, Saigal S, Willan AR. Planned caesarean section versus planned vaginal birth for breech presentation at term: a randomised multicentre trial. Term Breech Trial Collaborative Group. Lancet. 2000 Oct 21;356(9239):1375-83. doi: 10.1016/s0140-6736(00)02840-3. PMID 11052579
- [Background] ACOG Committee on Obstetric Practice. ACOG Committee Opinion No. 340. Mode of term singleton breech delivery. Obstet Gynecol. 2006 Jul;108(1):235-7. doi: 10.1097/00006250-200607000-00058. PMID 16816088
- [Background] Fok WY, Chan LW, Leung TY, Lau TK. Maternal experience of pain during external cephalic version at term. Acta Obstet Gynecol Scand. 2005 Aug;84(8):748-51. doi: 10.1111/j.0001-6349.2005.00505.x. PMID 16026399
- [Background] Lavoie A, Guay J. Anesthetic dose neuraxial blockade increases the success rate of external fetal version: a meta-analysis. Can J Anaesth. 2010 May;57(5):408-14. doi: 10.1007/s12630-010-9278-4. Epub 2010 Feb 3. PMID 20127530
- [Background] Weiniger CF, Ginosar Y, Elchalal U, Sharon E, Nokrian M, Ezra Y. External cephalic version for breech presentation with or without spinal analgesia in nulliparous women at term: a randomized controlled trial. Obstet Gynecol. 2007 Dec;110(6):1343-50. doi: 10.1097/01.AOG.0000295605.38175.7b. PMID 18055730
- [Background] Likis FE, Andrews JC, Collins MR, Lewis RM, Seroogy JJ, Starr SA, Walden RR, McPheeters ML. Nitrous oxide for the management of labor pain: a systematic review. Anesth Analg. 2014 Jan;118(1):153-67. doi: 10.1213/ANE.0b013e3182a7f73c. PMID 24356165
- [Background] Rosen MA. Nitrous oxide for relief of labor pain: a systematic review. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S110-26. doi: 10.1067/mob.2002.121259. PMID 12011877
- [Background] Creeley CE, Olney JW. The young: neuroapoptosis induced by anesthetics and what to do about it. Anesth Analg. 2010 Feb 1;110(2):442-8. doi: 10.1213/ANE.0b013e3181c6b9ca. Epub 2009 Dec 2. PMID 19955510
- [Background] Jevtovic-Todorovic V, Hartman RE, Izumi Y, Benshoff ND, Dikranian K, Zorumski CF, Olney JW, Wozniak DF. Early exposure to common anesthetic agents causes widespread neurodegeneration in the developing rat brain and persistent learning deficits. J Neurosci. 2003 Feb 1;23(3):876-82. doi: 10.1523/JNEUROSCI.23-03-00876.2003. PMID 12574416
- [Background] Schnabel A, Hahn N, Broscheit J, Muellenbach RM, Rieger L, Roewer N, Kranke P. Remifentanil for labour analgesia: a meta-analysis of randomised controlled trials. Eur J Anaesthesiol. 2012 Apr;29(4):177-85. doi: 10.1097/EJA.0b013e32834fc260. PMID 22273829
- [Background] Munoz H, Guerra S, Perez-Vaquero P, Valero Martinez C, Aizpuru F, Lopez-Picado A. Remifentanil versus placebo for analgesia during external cephalic version: a randomised clinical trial. Int J Obstet Anesth. 2014 Feb;23(1):52-7. doi: 10.1016/j.ijoa.2013.07.006. Epub 2014 Jan 3. PMID 24388737
- See also: ACOG committee opinion 340 — http://vb3lk7eb4t.search.serialssolutions.com.libproxy.lib.unc.edu/?sid=Entrez:PubMed&id=pmid:16816088
- See also: Neuraxial for version — https://link.springer.com/content/pdf/10.1007%2Fs12630-010-9278-4.pdf
- See also: Neuraxial for version — http://vb3lk7eb4t.search.serialssolutions.com.libproxy.lib.unc.edu/?sid=Entrez:PubMed&id=pmid:18055730
- See also: Nitrous for labor pain — http://vb3lk7eb4t.search.serialssolutions.com.libproxy.lib.unc.edu/?sid=Entrez:PubMed&id=pmid:24356165
- See also: nitrous for labor pain — https://ac-els-cdn-com.libproxy.lib.unc.edu/S0002937802701889/1-s2.0-S0002937802701889-main.pdf?_tid=8eaf7750-48b0-40b9-8efb-3085703ef78e&acdnat=1523306408_60b9557e881b9e75104aa6db52afedc9
- See also: Neuroapoptosis — http://vb3lk7eb4t.search.serialssolutions.com.libproxy.lib.unc.edu/?sid=Entrez:PubMed&id=pmid:19955510
- See also: anesthetic gases and apoptosis — http://www.jneurosci.org/content/jneuro/23/3/876.full.pdf
- See also: remi for labor analgesia — http://vb3lk7eb4t.search.serialssolutions.com.libproxy.lib.unc.edu/?sid=Entrez:PubMed&id=pmid:22273829

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitrous Oxide | Oxygen
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrous Oxide | Oxygen | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (4.7) | 31.8 (4.3) | 32.1 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 17 | 33
  Black/African American | 2 | 3 | 5
  Hispanic | 2 | 2 | 4
  Asian | 3 | 2 | 5
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48
Baby Weight [Mean (Standard Deviation); unit: Grams] — Newborn weight at time of delivery
  Grams | 3631.8 (491.2) | 3242.4 (416.6) | 3433.1 (491)
Amniotic Fluid Index (AFI) [Mean (Standard Deviation); unit: centimeters (cm)] — AFI is determined using ultrasound to measure the deepest vertical pocket of fluid in each quadrant. The four measurements are then added to calculate the AFI in cm. AFI between 8-18cm is considered normal. AFI < 5-6cm is considered low. AFI > 24-25cm is considered excessive. AFI > 10cm has been shown to be associated with successful ECV.
  centimeters (cm) | 12.3 (4.5) | 11.1 (4.2) | 11.6 (4.3)
Gestational Age [Median (Standard Deviation); unit: Weeks] — Gestational age of the patient at the time of version procedure.
  Weeks | 37.1 (0.4) | 37.2 (0.4) | 37.1 (0.4)
BMI [Mean (Standard Deviation); unit: Kg/m^2] — Basal Metabolic Rate
  Kg/m^2 | 29.3 (5.1) | 31 (6.3) | 30.2 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Score Experienced During Version
Description: Pain scores will be collected following each version attempt using an 11 point scale (with 0 being no pain at all; 10 being worst pain imaginable), ranging from 0 to 10. Higher scores indicate more pain, lower scores indicate less pain. If more than one attempt, pain scores will be averaged to obtain a single score for the entire procedure.
Time Frame: During each version procedure, a total average of up to approximately 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nitrous Oxide | Oxygen
Number analyzed (Participants) | 24 | 24
score on a scale | 5.486 (2.307) | 5.433 (2.695)
Statistical Analysis 1: Comparison: Nitrous Oxide vs Oxygen; Test type: Equivalence — The equivalence margin is the standard error of the estimated difference; p = 0.943, t-test, 2 sided; Mean Difference (Final Values) = 0.053, 95% CI 2-sided [-1.402 to 1.507], Standard Deviation 2.508

2. Secondary Outcome: Mean Anxiety Score Experienced During Version
Description: Anxiety scores will be collected following each version attempt using an 11 point scale (0 being not at all anxious; 10 being extremely anxious), ranging from 0 to 10. Higher scores indicate more anxiety, lower scores indicate less anxiety. If more than one attempt, anxiety scores will be averaged to obtain a single score for the entire procedure.
Time Frame: During each version procedure, a total average of up to approximately 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nitrous Oxide | Oxygen
Number analyzed (Participants) | 24 | 24
score on a scale | 4.696 (2.969) | 4.253 (2.762)
Statistical Analysis 1: Comparison: Nitrous Oxide vs Oxygen; Test type: Equivalence — The equivalence margin is the standard error of the estimated difference; p = 0.597, t-test, 2 sided; Mean Difference (Final Values) = 0.443, 95% CI 2-sided [-1.229 to 2.114], Standard Deviation 2.867

3. Secondary Outcome: Mean Post-procedure Pain Score
Description: Pain scores will be collected following completion of the version using an 11 point scale (0 being no pain at all; 10 being worst pain imaginable), ranging from 0 to 10. Higher scores indicate more pain, lower scores indicate less pain.
Time Frame: Immediately Post-procedure, within approximately 15 minutes of final version attempt
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nitrous Oxide | Oxygen
Number analyzed (Participants) | 24 | 24
score on a scale | 1 (1.155) | 0.88 (1.394)
Statistical Analysis 1: Comparison: Nitrous Oxide vs Oxygen; Test type: Equivalence — The equivalence margin is the standard error of the estimated difference; p = 0.748, t-test, 2 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.629 to 0.869], Standard Deviation 1.280

4. Secondary Outcome: Mean Post-procedure Patient Satisfaction Score
Description: Satisfaction will be assessed following the procedure using an 11 point scale (0 being not at all satisfied; 10 being extremely satisfied), ranging from 0 to 10. Higher scores indicate more satisfaction, lower scores indicate less satisfaction.
Time Frame: Immediately Post-procedure, within approximately 15 minutes of final version attempt
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nitrous Oxide | Oxygen
Number analyzed (Participants) | 24 | 24
score on a scale | 4.286 (4.027) | 6.920 (3.593)
Statistical Analysis 1: Comparison: Nitrous Oxide vs Oxygen; Test type: Equivalence — The equivalence margin is the standard error of the estimated difference; p = 0.025, t-test, 2 sided; Mean Difference (Final Values) = -2.634, 95% CI 2-sided [-4.927 to -0.341], Standard Deviation 3.816

5. Secondary Outcome: Mean Post-procedure Provider Assessed Level of Difficulty Score
Description: Following the procedure, the obstetric provider performing the procedure will rate the ease of procedure on a 1-10 scale (1 being very easy and 10 being extremely difficult), ranging from 1 to 10. Higher scores indicate more difficulty, lower scores indicate less difficulty. A 10 point scale was used for this outcome, while an 11 point scale was used for the other 4 outcome measures (pain, anxiety, post-procedure pain and satisfaction).
Time Frame: Immediately Post-procedure, within approximately 15 minutes of final version attempt
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nitrous Oxide | Oxygen
Number analyzed (Participants) | 24 | 24
score on a scale | 6.136 (2.21) | 6.080 (3.187)
Statistical Analysis 1: Comparison: Nitrous Oxide vs Oxygen; Test type: Equivalence — The equivalence margin is the standard error of the estimated difference; p = 0.944, t-test, 2 sided; Mean Difference (Final Values) = 0.056, 95% CI 2-sided [-1.543 to 1.655], Standard Deviation 2.742

ADVERSE EVENTS:
Time Frame: During each version procedure (or attempt), a total average of up to approximately 30 minutes and through approximately 15 minutes post-procedure following the final version attempt.
Arm/Group | Nitrous Oxide | Oxygen
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 5/24 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nitrous Oxide (N=24) | Oxygen (N=24)
Nausea (Gastrointestinal disorders) | 2 | 2
Transient headache (General disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT03502915/Prot_SAP_000.pdf